CLINICAL TRIAL: NCT03906292
Title: Frontline Asciminib Combination in Chronic Phase CML
Acronym: CMLXI
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Jena (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other); Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Thomas Ernst, PD Dr. med., Principal Investigator, University of Jena
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fascination; 2024-516212-24-00 (EU CTIS Number)
Record Dates: First submitted 2018-12-14; First posted 2019-04-08 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate; asciminib; nilotinib; BID protein, human; Dasatinib

STUDY DESIGN:
Intervention Model Description: 5 parallel cohorts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Asciminib 60mg QD (Experimental): Standard therapy of Imatinib 400 mg QD and asciminib 60 mg QD
  Interventions: Drug: Imatinib; Drug: Asciminib
- Asciminb 20 mg BID (Experimental): Standard therapy of Nilotinib 300 mg BID and asciminib 20 mg BID
  Interventions: Drug: Nilotinib 300 mg; Drug: Asciminib
- Asciminib 40 mg QD (Experimental): Standard therapy of Nilotinib 300 mg BID and asciminib 40 mg QD
  Interventions: Drug: Nilotinib 300 mg; Drug: Asciminib
- Asciminib 80 mg QD (Experimental): Standard therapy of Dasatinib 100 mg QD and asciminib 80 mg QD
  Interventions: Drug: Dasatinib; Drug: Asciminib
- Asciminib 80 mg QD monotherapy (Experimental): Asciminib 80 mg QD as a single agent
  Interventions: Drug: Asciminib

INTERVENTIONS:
Drug: Imatinib — Imatinib 400 mg QD and asciminib 60 mg QD
  Other Names: Imatinib 400 mg QD and asciminib 60 mg QD
  Arms: Asciminib 60mg QD
Drug: Nilotinib 300 mg — Nilotinib 300 mg BID and asciminib 20 mg BID or 40 mg QD
  Other Names: Nilotinib 300 mg BID and asciminib 20 mg BID or 40 mg QD
  Arms: Asciminb 20 mg BID; Asciminib 40 mg QD
Drug: Dasatinib — Dasatinib 100 mg QD and asciminib 80 mg QD
  Other Names: Dasatinib 100 mg QD and asciminib 80 mg QD
  Arms: Asciminib 80 mg QD
Drug: Asciminib — Asciminib 80 mg QD Monotherapy

SUMMARY:
Adult male and female patients with newly diagnosed Philadelphia chromosome positive (Ph+) and/or BCR-ABL1 positive CML can be included in the study until 3 months after diagnosis. A <4 week pretreatment with hydroxyurea is permitted. Patients treated for <6 weeks with nilotinib 300 mg BID, imatinib 400 mg QD, dasatinib 100 mg QD or without any therapy are eligible for recruitment and will be allocated to the respective cohort. All patients must provide written informed consent to be enrolled in the trial. Cohorts were designed to allow assessment of QD and BID asciminib based combinations to optimize quality of life and compliance. Patients will not be randomized. In general, cohorts will be filled consecutively. Asciminib therapy will be commenced 12 weeks after start of nilotinib, imatinib or dasatinib and after recovery of hematopoiesis or in case of no therapy so far 6 weeks after diagnosis as first line treatment. Referred patients already treated with imatinib, nilotinib or dasatinib will remain on the initial drug and will be allocated to the respective cohort.

DETAILED DESCRIPTION:
Despite the dramatic progress made over the past decade with TKIs in the treatment of CML, allogeneic stem cell transplant remains the only proven curative therapy. To achieve cure or benefit from treatment-free remissions with pharmacologically-based therapies, it is estimated that patients will likely need to achieve a sustained reduction in tumor burden corresponding to a deep molecular response of at least 4 logs (MR4). Currently, only 30.8% of patients achieve a deep molecular response after 12 months of treatment with single agent nilotinib.

The development of the novel and potent BCR-ABL1 allosteric inhibitor, asciminib, presents an opportunity to assess the effect of a different mechanism of inhibition of BCR-ABL1 in the first-line treatment of CML to enhance speed of response and to increase the patient population benefitting from deep molecular response. Dosing a combination of asciminib with an ATP-site inhibitor also has the potential to prevent the emergence of resistance due to point mutations being acquired in one of the binding sites.

The safety, tolerability and pharmacokinetic profile of asciminib as a single agent and in combination with either nilotinib or imatinib or dasatinib was assessed in a phase-I study. At the doses chosen here, all three combination treatments were well tolerated.

Since in all patient cohorts the standard of care therapy will remain the backbone of initial therapy, there is no reason to expect an efficacy problem with the combination therapies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with diagnosis of CP-CML with cytogenetic confirmation of the Ph+ chromosome [t(9;22)(q34;q11)].
* Ph-negative cases or patients with variant translocations who are BCR-ABL1 positive in multiplex PCR 35 will be also considered eligible.
* ECOG performance status of ≤2.
* Age ≥ 18 years old (no upper age limit is given)
* Serum levels of potassium, magnesium, total calcium within the normal limits (≥LLN [lower limit of normal] and ≤ULN [upper limit of normal]). Correction of electrolytes levels with supplements to fulfil enrolment criteria is allowed.
* AST and ALT ≤2.5 x ULN or 5.0 x ULN if considered due to leukemia
* Alkaline phosphatase ≤2.5 x ULN unless considered due to leukemia
* Total bilirubin ≤1.5 x ULN, except known Gilbert disease
* Serum creatinine ≤2 x ULN
* Written informed consent prior to any study procedures being performed.

Exclusion Criteria:

* Allogeneic stem cell transplantation
* Known impaired cardiac function, including any of the following:

  * Congenital long QT syndrome
  * History of or presence of clinically significant ventricular or atrial tachyarrhythmia
  * QTc >450 msec on screening ECG
  * Myocardial infarction within 12 months prior to starting therapy
* Other clinical significant heart disease (e.g. unstable angina, congestive heart failure)
* Acute or chronic viral hepatitis with moderate or severe hepatic impairment (Child-Pugh scores >6), even if controlled
* Other concurrent uncontrolled medical conditions (e.g., active or uncontrolled infections, acute or chronic liver and renal disease) that could cause unacceptable safety risks or compromise compliance with the protocol
* Impaired gastrointestinal function or disease that may alter the absorption of study drug (e.g., ulcerative disease, uncontrolled nausea, vomiting and diarrhea, malabsorption syndrome, small bowel resection or gastric by-pass surgery)
* Concomitant medications known to be strong inducers or inhibitors of the CYP450 isoenzyme CYP3A4
* Patients who have undergone major surgery ≤2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Patients who are pregnant or breastfeeding or women of reproductive potential not employing an effective method of birth control. Women of childbearing potential must have a negative serum pregnancy test within 14 days of study start. Post-menopausal women must be amenorrheic for at least 12 months in order to be considered of non-childbearing potential. Male and female patients must agree to employ an effective method of birth control throughout the study and for up to 2 weeks following discontinuation of study drug
* Known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory)
* Known serious hypersensitivity reactions to asciminib, imatinib, nilotinib or dasatinib
* Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention
* Patients unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
deep molecular response (Rate of MR4) | at month 12 after Start of Standard-Therapy
  Achievement of deep molecular response (MR4) throught standardized testing of BCR-ABL-transcript Levels
deep molecular Response (Rate of MR4.5) | at month 36 after Start of Standard-Therapy
  Achievement of deep molecular response (MR4.5) throught standardized testing of BCR-ABL-transcript Levels

SECONDARY OUTCOMES:
molecular response (MMR and MR4.5) | at and by 6, 12, 18, 24, 36 and 60 months after Start of Therapy
  Achievement of deep molecular response throught standardized testing of BCR-ABL-transcript levels
Adverse Events | at and by baseline, 3, 6, 12, 15, 18, 21, 24, 36 and 60 months after Start of Therapy
  Incidence of adverse events grade 1-5 and 3-5
Progression free survival | at month 60 after Start of Therapy
  Progression free survival at the end of the study
Overall survival | at month 60 after Start of Therapy
  Overall survival at the end of the study
Maintenance of MR4.5 during Asciminib-monotherapy | at month 36 and 60 after Start of Therapy
  Achievement of deep molecular response (MR4.5) throught standardized testing of BCR-ABL-transcript Levels
Achievement and durability of treatment-free remission | months 37 and 60 after Start of Therapy
  Achievement of deep molecular response (MR4) throught standardized testing of BCR-ABL-transcript Levels

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ernst, Prof. Dr., Principal Investigator — University Hospital Jena
Locations (21):
- Germany (21):
  - Universitätsklinikum Aachen Medizinische Klinik IV, Aachen
  - Charite Universitätsmeditin Berlin, Campus Virchow Klinikum, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Klinikum Bremen Mitte, Bremen
  - Klinikum Chemnitz gGmbH, Chemnitz
  - GOKOS GmbH, Dresden
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Dresden
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Leipzig, Leipzig
  - Gemeinschaftspraxis Dres. Müller/ Kröning/ Jentsch-Ullrich/ Tietze/ Krogel, Magdeburg
  - Universitätsmedizin der Johannes- Gutenberg Universität Mainz, Mainz
  - Universitätsmedizin Mannheim, Mannheim
  - Universitätsklinikum Gießen und Marburg, Marburg
  - Klinikum rechts der Isar, München
  - Brüderkrankenhaus St. Josef Paderborn, Paderborn
  - Krankenhaus Barmherzige Brüder Regensburg, Regensburg
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No